CLINICAL TRIAL: NCT01566708
Title: Diagnostic and Interventional Study of Neuro-Music Therapy for Recent Onset Tinnitus: Evaluation of a Therapy Concept Using Psychological Assessment and Functional Neuroimaging
Brief Title: Neuro-Music Therapy for Recent Onset Tinnitus: Evaluation of a Therapy Concept
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: German Center for Music Therapy Research (Other)
Collaborators: Heidelberg University (Other); Clinic of Diagnostic and Interventional Neuroradiology, Saarland University Clinic, Homburg, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMTR-TA-01; 00.181.2011 (Other Grant/Funding Number: Klaus Tschira Foundation (KTF))
Record Dates: First submitted 2012-03-23; First posted 2012-03-29 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Tinnitus
Keywords: Acute Tinnitus; Recent Onset Tinnitus; Music Therapy; fMRI; Therapy Evaluation
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- treatment group (Experimental)
  Interventions: Behavioral: Neuro-Music Therapy immediately
- waiting list group (Active Comparator)
  Interventions: Behavioral: Neuro-Music Therapy after waiting time
- control group (Active Comparator)
  Interventions: Behavioral: Music-therapeutical stress management coaching

INTERVENTIONS:
Behavioral: Neuro-Music Therapy immediately — 20 patients are randomized to receive Neuro-Music Therapy immediately. Neuro-Music Therapy takes 5 days and comprises 9 consecutive 50-minutes sessions of individual therapy. Immediately before and after treatment extensive diagnostics are performed, including psychological assessment, functional neuroimaging and electro-physiological examinations.
  Arms: treatment group
Behavioral: Neuro-Music Therapy after waiting time — 20 Patients were randomized to receive Neuro-Music Therapy after a waiting period not exceeding 6 weeks. Within this waiting time, patients undergo exactly the same diagnostic procedure as the patients of the treatment group.
  Arms: waiting list group
Behavioral: Music-therapeutical stress management coaching — 20 non-tinnitus controls matched in age, gender and hearing ability receive a music-therapeutical stress coaching program. This intervention is based on the main treatment components of the Neuro-Music Therapy for acute tinnitus with alterations of the tinnitus specific elements. Immediately before and after this five-day coaching, controls undergo exactly the same diagnostic procedure as the patients of the treatment group.
  Arms: control group

SUMMARY:
To date, the pharmacological treatment options for tinnitus are unsatisfactory. For acute tinnitus drug treatments are only rated as being successful in approximately half of all cases. Therefore, the purpose of this study is to evaluate a neuro-music therapeutic approach (the "Heidelberg Model of Music Therapy") as a new treatment option for patients with recent onset tinnitus after initial medical treatment has failed.

DETAILED DESCRIPTION:
Acute tinnitus is the phenomenon of ringing or buzzing in the ears without an external sound source that is persisting for a maximum of three month. Several pharmacological treatment options for acute tinnitus have been established. Nonetheless, after initial medical intervention, tinnitus symptoms are often persisting and leading to substantial distress.

The objective of the present study is to examine the efficacy of the "Heidelberg Model of Music Therapy" for patients with recent onset tinnitus whose tinnitus symptoms are enduring after pharmacological treatment. The "Heidelberg Model of Music Therapy" is a manualized short term music therapeutic intervention lasting for 9 consecutive 50-minutes sessions of individualized therapy. It strives for an integration of strategies to manage the psychological state and possibly restore the underlying neurophysiological reorganisation. At the basis of this music therapy concept is the notion that tinnitus is experienced as an auditory percept - just as musical stimuli are experienced as auditory percepts. An outstanding feature of this treatment approach is the way in which patients actively influence their symptoms. This leads to an improved self-efficacy and a more differentiated picture of their symptomatology.

For patients with chronic subjective tinnitus the "Heidelberg Model of Music Therapy" has proven to be an efficient means to reduce tinnitus distress and loudness. Prior studies indicate that these positive results are due to the beneficial influence of the music therapy on the neuronal structures underlying tinnitus pathology.

In the present study the effects of the music therapeutic intervention on tinnitus severity and tinnitus distress for patients with acute tinnitus are evaluated on the basis of a battery of psychological tests as well as psycho-physiological measurements. A task-based functional magnetic resonance imaging (fMRI) paradigm is used to investigate alterations in neuronal networks supposed to be involved in tinnitus perception and chronification.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute tinnitus persisting for a maximum of 3 month
* Adults, aged 18 or over
* No contraindication for MRI scan
* Initial medical intervention is accomplished
* Patients are able to understand, read and speak German fluently
* Patients are able to give written informed consent

Exclusion Criteria:

* Clinical diagnosis of chronic tinnitus persisting for longer than 3 month
* Tinnitus related to anatomic lesions of the ear, to retrocochlear lesions or to cochlear implantation
* Clinical diagnosis of severe mental disorder
* Clinical diagnosis of Menière's Disease
* Severe hyperacusis
* Severe hearing impairment
* Any contraindication for MRI scan
* Initial medical intervention is not accomplished
* Patients are not able to understand, read and speak German fluently
* Patients are not able to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Questionnaire (TQ, Goebel and Hiller 1998) total score change from baseline to end of treatment | baseline to week 1 and 12
Tinnitus-Beeinträchtigungs-Fragebogen (TBF-12, Greimel et al. 2000) total score change from baseline to end of treatment | baseline to week 1 and 12

SECONDARY OUTCOMES:
change in tinnitus frequency | baseline to day 1, 2, 3 and 4 of treatment
change in electro-physiological variables (skin temperature, skin conductance level, pulse frequency, respiration frequency) | baseline to day 1, 2, 3, 4 and 5 of treatment
task-based fMRI: change in neuronal activity from baseline to end of treatment | baseline to week 1
Attention and Performance Self Assessment Scale (APSA, Görtelmeyer et al. 2012) total score change from baseline to end of treatment | baseline to week 1 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Hans V Bolay, Prof. Dr., Study Director — German Center for Music Therapy Research; Miriam Grapp, Principal Investigator — German Center for Music Therapy Research
Locations (1):
- German Center for Music Therapy Research, Heidelberg, Baden-Wurttemberg, Germany